CLINICAL TRIAL: NCT01103297
Title: A Prospective Multicenter Case-series of Patients Treated With the 2.4 mm Variable Angle LCP Two-Column Volar Distal Radius Plate ®
Brief Title: 2.4 mm Variable Angle LCP Two-Column Volar Distal Radius
Acronym: VALCP2010
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VALCPDR
Record Dates: First submitted 2010-03-25; First posted 2010-04-14 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Distal Radius Fractures
Keywords: Distal radius fracture; Double row plate; Volar approach; DVR plate; Postoperative complications [MeSH]
MeSH Terms: conditions — Wrist Fractures | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Variable Angle Distal Radius Plate (Other)
  Interventions: Device: Variable Angle Distal Radius Plate ® (Surgery)

INTERVENTIONS:
Device: Variable Angle Distal Radius Plate ® (Surgery) — Fracture reduction with distal radius plate
  Other Names: 2.4 Variable Angle LCP Two-Column Volar Distal Radius Plate®

SUMMARY:
The purpose of this study is to is to evaluate the postoperative loss of reduction rate in patients with distal radius fractures treated using the 2.4 mm Variable Angle LCP Two-Column Volar Distal Radius Plate ®.

DETAILED DESCRIPTION:
The treatment of choice for distal radius fractures is anatomic reduction with stable fixation. This is commonly achieved via open reduction and internal fixation with angle-stable designed locking plates using either a volar or dorsal approach. Frequent complications of tendinitis are associated with the latter approach. Palmar application of angle-stable plates reduces this problem of extensor tendon irritation; however a high incidence of fracture collapse has been documented. Currently, there are no existing locking plates that provide sufficient stability particularly for complex fractures. Insufficient fragment fixation can result in loss of reduction due to interfragmentary movement and lead to mal- or nonunion.

The Variable Angle LCP Two-Column Volar DR plate (VA LCP DR) is a novel development of the LCP Distal Radius Plate System, which is designed to treat a wide variety of distal radius fracture patterns. Because of its design (ie, low plate and screw profile, polished surface, rounded edges, various locking options), not only can the potential for tendon adhesions and soft tissue irritation be minimized, the plate can address fragments individually for each fracture type. Thus, the versatility of VA LCP facilitates the reduction and stabilization of even the most complex fractures, including those in osteoporotic bone.

This prospective case-series will evaluate the performance of the new VA LCP DR plate in the treatment of complex articular fractures of the distal radius. The primary objective of this study involves the documentation of postoperative loss of reduction; functional outcomes, quality of life and rate of complications associated with fracture fixation will also be assessed as part of the secondary study aims.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Patients with closed, partial or complete articular distal radius fractures classified as: AO 23 B3 and AO 23 C1, C2, C3 confirmed by CT scan
* Definitive primary fracture treatment with a VA LCP DR
* The patient is willing and able to participate in the study follow-up examinations according to the protocol
* The patient is able to understand and read the local language at an elementary level
* The patient or his/her legal guardian is willing and able to give his informed consent to participate in the study
* Woman must be one of the following:
* Postmenopausal defined as amenorrhea for at least 6 months before screening and a serum follicle stimulating hormone (FSH) level consistent with postmenopausal status
* Surgically sterile, (have had a hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy)
* Abstinent (at the discretion of the investigator) or,
* If sexually active, be practicing an effective method of birth control such as hormonal prescription oral contraceptives, progesterone implants or injections, intrauterine device (IUD), a double-barrier method such as condoms, diaphragms or cervical caps with spermicidal foam, cream or gel, or male partner with a vasectomy.
* Women of childbearing potential must have a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test, or a negative urine pregnancy test at screening.

Exclusion Criteria:

* Previous ipsilateral distal radius fracture
* Other fractures of the ipsilateral side (except ulna)
* Pathologic fracture due to malignancy
* The patient suffers from a polytrauma
* The patient is affected by drug or alcohol abuse
* The patient suffers from active malignancy
* Neurological and psychiatric disorders
* The patient has participated in any other device or drug related clinical trial within the previous month
* The patient is a prisoner
* Breast feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2010-06; Primary Completion 2014-02 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Loss of reduction | over 1 year
  Loss of reduction will be defined as the change in measurement* determined to 0.5 mm or 1 degree of accuracy:
  *Any change in angles, length or secondary fragment displacement (ie, radial height (length), radial inclination, ulnar variance, gap, step-off, palmar tilt (inclination) / dorsal tilt, scapholunate angle, teardrop angle, and the AP distance).

SECONDARY OUTCOMES:
Rate of fracture fixation complications | Baseline
Wrist function | 12 weeks
  Bilateral Range of motion (ROM)
Grip strength | 12 weeks
  With Jamar dynamometer
Wrist pain and disability in functional activities | Baseline
  Patient self-assessment of wrist function questionnaire (PRWE)
Quality of Life | Baseline
  Health-related quality of life (EQ5D)
Implantation and system feedback | Baseline
Rate of fracture fixation complications | 12 weeks
Rate of fracture fixation complications | 1 year
Wrist function | 1 year
  Bilateral Range of motion (ROM)
Grip strength | 1 year
  With Jamar dynamometer
Wrist pain and disability in functional activities | 12 weeks
  Patient self-assessment of wrist function questionnaire (PRWE)
Wrist pain and disability in functional activities | 1 year
  Patient self-assessment of wrist function questionnaire (PRWE)
Quality of Life | 12 weeks
  Health-related quality of life (EQ5D)
Quality of Life | 1 year
  Health-related quality of life (EQ5D)

CONTACTS AND LOCATIONS:
Overall Officials: Jesse B Jupiter, MD, Principal Investigator — Massachusetts General Hospital, Orthopaedic Surgery, Yawkey Center, Suite 2100, 55 Fruit Street, Boston, MA 02114, USA; Andreas Schierz, MD, Principal Investigator — Spital Zollikerberg, Unfallchirurgie, Trichtenhauserstrasse 20, CH-8125 Zollikerberg, Switzerland
Locations (6):
- Unfallkrankenhaus Graz, Graz, Austria
- Germany (2):
  - Charite Berlin, Berlin
  - Universitätssklinikum Münster, Münster
- Switzerland (3):
  - Universitätsspital Basel, Basel, Basel
  - Luzerner Kantonsspital, Lucerne, Canton of Lucerne
  - Spital Zollikerberg, Zurich